CLINICAL TRIAL: NCT05351632
Title: Clinical Validation and Evaluation of Reliability of Comprehensive Complication Index (CCI) for Recording Percutaneous Nephrolithotomy Complications
Brief Title: Comprehensive Complication Index in the Classification of Complications of Percutaneous Nephrolithotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Collaborators: Zonguldak Bulent Ecevit University (Other); Ankara University (Other); Inonu University (Other); Istanbul University (Other); Acibadem University (Other); Eskisehir Osmangazi University (Other); Başakşehir Çam & Sakura City Hospital (Other Government); Koç University (Other); Izmir Metropolitan Municipality Esrefpasa Hospital (Unknown); Alanya Alaaddin Keykubat University (Other); Cukurova University (Other); Ondokuz Mayıs University (Other); Dokuz Eylul University (Other); Samsun Education and Research Hospital (Other); Gazi University (Other); Hacettepe University (Other); Abant Izzet Baysal University (Other); Ankara Training and Research Hospital (Other); Hitit University (Other); Baskent University (Other)
Responsible Party: Principal Investigator, Yiloren Tanidir, Associ.Prof., Marmara University
Other Study IDs: 2022/06-7
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Complications, Postoperative
Keywords: Comprehensive Complications Index; Percutaneous Nephrolithotomy; Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative complications should be reported systematically, objectively and reproducibly. The Clavien-Dindo Classification (CDC), first described in 2004, is the most popular classification system still in use today for assessing perioperative morbidity and mortality. In 2018, the European Association of Urology (EAU) validated this classification, which was originally defined for general surgery operations, for urological operations as well. There are aspects of the CDC that can be critical and weak. The CDC's main weakness is that in the vast majority of studies it only considers the most serious complications. Minor complications are often overlooked and the overall complication burden is therefore underestimated. Because of this vulnerability, it is difficult to compare complications from different patients. For example, it cannot be determined whether a patient with two Grade I complications has higher postoperative morbidity than a patient with one Grade II complication. To address these limitations, the Comprehensive Complications Index (CCI) was defined in 2013 as a new and more comprehensive scoring system for surgical complications.

The CCI is essentially an index based on the CDC, but sums all postoperative complications by severity and scores them on an interval scale. It is scored from 0 (no complications) to 100 (patient's death) for each patient.

CCI in Urology Practice; Validated for Radical Cystectomy, Radical Prostatectomy, Radical Nephroureterectomy, Partial Nephrectomy.

In recent years, validation studies of this index have been carried out in endourological surgeries.

DETAILED DESCRIPTION:
Percutaneous kidney stone surgery (PNL) will be performed due to kidney stones, and 644 patients will be included in the study according to the power analysis*. Demographic data of the patients, stone characteristics and data related to stone burden, data related to the operation will be noted by looking at the hospital files. Patients who have undergone surgery can be discharged after an average of 3 days and can be called for routine control after an average of 2 months. All complications developed during the inpatient follow-up and any complications developed during the control period will be noted using the patient's file information. Then, all these complications that are detected to develop will be scored separately using the CCI and CDC complication scales.

1. Using the free online tool www.assessurgery.com, the Comprehensive Complications Index (CCI) score for the total burden of complications will be calculated for each patient.
2. Each patient's most major complication will be determined and graded according to the Clavien-Dindo (CDC) classification (as described below).

Grade I: Any deviation from the normal postoperative course requiring only the following drugs: antiemetics, antipyretics, diuretics Grade II: Pharmacological therapy (with drugs not necessary for CDC I complications), blood transfusion, total parenteral nutrition Grade IIIa: Surgical, endoscopic or radiological intervention not under general anesthesia Grade IIIb: Surgical, endoscopic or radiological intervention under general anesthesia Grade IVa: single organ dysfunction requiring intensive care unit management Grade IVb: multiple organ dysfunction requiring intensive care unit management Grade V: Death

All the data obtained, CCI and CDC, will be compared among themselves in terms of reliability, demographic data obtained from the pre-operative file data, stone characteristics and data related to the operation will be compared, as well as their relationship with the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* To have a medical indication for percutaneous kidney stone surgery
* To have given consent to participate in the study
* To be18 years of age or older

Exclusion Criteria:

* To be under the age of 18
* Not to have given consent to participate in the study
* Not to have a medical indication for percutaneous kidney stone surgery
* To Have an orthopedic disorder that prevents him from undergoing percutaneous kidney stone surgery
* To have a hematological disorder that prevents percutaneous kidney stone surgery
* To have a malignancy that prevents percutaneous kidney stone surgery
* To have a serious cardiac and respiratory comorbidities that prevent percutaneous kidney stone surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient group over 18 years of age with kidney stones and no contraindications for PCNL
Sampling Method: Non-Probability Sample
Enrollment: 644 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The Comprehensive Complication Index | within 2 months post-procedure
  The comprehensive complications index was proposed as a novel comprehensive scoring system for surgical complications in 2013. It's scoring complications on an interval scale between 0 (no complication) and 100 (death of the patient) for each patient.
Clavien-Dindo-Classification score | within 2 months post-procedure
  The Clavien-Dindo-Classification (CDC), first described in 2004, is the most popular classification system for assessing perioperative morbidity and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Reha GİRGİN, Assist.Prof., Study Director — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bülent Ecevit University, school of medicine, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No